CLINICAL TRIAL: NCT02775955
Title: A Phase-1 Study Comparing the Pharmacokinetics of Intranasal RX0041-002 in Subjects With Severe Renal Impairment and Subjects With Normal Renal Function
Brief Title: PK Study of Intranasal RX0041-002 in Subjects With Severe Renal Impairment and Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Project Solutions, Inc. (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTS2015013
Record Dates: First submitted 2016-03-23; First posted 2016-05-18 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — FG 0041

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RX0041-002 (Experimental): Active
  Interventions: Drug: RX0041

INTERVENTIONS:
Drug: RX0041 — Active
  Other Names: 0041

SUMMARY:
The primary objective of this study is to evaluate the potential effect of renal impairment on the systemic pharmacokinetics of acute Intranasal RX0041-002. The secondary objective is to evaluate the safety and tolerability of acute Intranasal RX0041-002 in subjects with normal renal function and severe renal impairment.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the potential effect of renal impairment on the systemic pharmacokinetics of acute Intranasal RX0041-002. The secondary objective is to evaluate the safety and tolerability of acute intranasal RX0041-002 in subjects with normal renal function and severe renal impairment.

2 INVESTIGATOR/STUDY SITE

The study will be conducted at Comprehensive Clinical Research in Berlin, New Jersey. The principal investigator will be Dr. David Hassman. Institutional review will be performed by Chesapeake Institutional Review Board..

3 BACKGROUND

Cocaine Hydrochloride Topical Solution (4%) is currently available for the induction of local (topical) anesthesia of accessible mucous membranes of the oral, laryngeal and nasal cavities (DESI product). Pennsylvania Pain Specialists (PPS) are seeking FDA approval for RX0041-002 as a topical anesthetic for diagnostic and surgical procedures in the nasal cavity.

Cocaine is a naturally-derived local anesthetic with a long history of use. Like other structurally-related local anesthetics, cocaine produces direct effects on cell membranes. Cocaine blocks sodium channel activity and thus prevents the generation and conduction of nerve impulses in electrically active cells. Cocaine also has vasoconstriction properties which for surgical or diagnostic procedures of the mucous membranes of the nasal cavities decreases operative bleeding and improves surgical visualization. The therapeutic use of cocaine hydrochloride, 4% solution topically applied to the nasal septum for local anesthesia is reported in the public clinical literature but has never received official FDA approval for this indication. It has been used in surgical procedures involving the nose, throat, larynx and lower respiratory passages because blood loss from these highly vascularized areas can be considerable and may also obscure the operative field.

The pharmacokinetics of cocaine administered via nasal absorption has been reported in the literature. However, regardless of the route of administration, several studies have shown that cocaine has a plasma half-life of 0.5-1.5 h, an apparent volume of distribution of 2-3 L/kg, and an apparent systemic clearance of ≈2 L/min. Only 1-5% of cocaine is cleared unmetabolized in urine, where it may be detected for only 3-6 h after use. The primary pathway of cocaine elimination is by hydrolysis of its two ester groups to form the two major inactive metabolites, ecgonine methyl ester (EME) and benzoylecgonine (BE), with half-lives of approximately 4 and 6 h, respectively. These compounds constitute over 80% of cocaine's metabolites and are detected in urine for 14-60 h after cocaine administration. Norcocaine, a minor but active metabolite, is formed by cytochrome P450 (CYP 3A4) mediated N-demethylation of cocaine. However, only 2% - 6% of cocaine is metabolized to norcocaine in humans.

The present study is being conducted to evaluate the potential effects of renal impairment on the pharmacokinetics of cocaine, its major metabolites and the active metabolite (norcocaine) after (4%) intranasal cocaine HCl topical administration, at the typical clinical dose of 160 mg.

4 SUMMARY OF DRUG INFORMATION

RX0041-002 (Cocaine HCl, USP) is a crystalline, granular, or powder substance having a saline, slightly bitter taste that numbs tongue and lips. Each mL of RX0041-002 Topical Solution contains Cocaine HCl 40 mg (4%) as an aqueous solution.

5 SUBJECT POPULATION

The subject population for this study will include male and female adults (≥ 18 years). A sufficient number of subjects will be enrolled to complete 8 subjects with severe renal impairment and 8 subjects with normal renal function. The subjects with normal renal function will be selected in order to match the subjects with renal impairment in terms of age, sex and BMI. For assignment to the treatment groups, severe renal impairment will be defined as an eGFR of 15-29 mL/min/1.73m2. Normal renal function will be defined as an eGFR ≥ 90 mL/min/1.73m2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Greater than or equal to 18 years of age and able to understand and comply with protocol requirements, provide written informed consent and HIPPA authorization; ± 10 years for individual age-matched controls.
3. Females (if of child-bearing potential and sexually active) and males (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method from the first dose and for 8 days following administration of study drug. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm, intrauterine device (IUD), condom, surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method or withdrawal.
4. BMI ≥ 18 ≤ 42 (see Appendix); ± 20% for BMI-matched controls
5. In general, good health aside from renal disease and associated conditions as ascertained by physical examination (PE) including measurement of supine and standing vital signs, medical history, clinical laboratory studies, and 12-lead electrocardiogram (ECG).
6. For assignment to the normal renal function (control) group, subjects must have an eGFR ≥ 90 mL/min/1.73m2 at screening. Assignment to the severe renal impairment group will be based upon an eGFR of 15-29 mL/min/1.73m2 at screening.
7. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance.

Exclusion Criteria:

1. Has a known allergy to any ester based anesthetics including cocaine HCl, procaine, tetracaine, chloroprocaine, dibucaine, or benzocaine amide based anesthetic allergies are NOT exclusionary. Amide based anesthetics are : lidocaine, mepivicaine, bupivicaine, levobupivicaine, ropivicaine, etidocaine, prilocaine, and articaine.
2. Concurrent use of medications known to affect the elimination of serum creatinine (eg, trimethoprim/sulfamethoxazole [Bactrim®] or cimetidine [Tagamet®]) and competitors of renal tubular secretion (eg, probenecid) within 30 days prior to the first dose of study drug.
3. Presence of significant gastrointestinal, liver or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
4. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study.
5. The use of amphetamines, methylphenidate or other stimulant prescription and nonprescription products such as pseudoephedrine, bronchial inhalers containing sympathomimetics (epinephrine or other beta-receptor agonist) or herbal products in the 7 days prior to screening or has a need to use these drugs during the course of the study.
6. Use of any selective serotonin and norepinephrine reuptake inhibitorsserotonin-specific reuptake inhibitors antidepressants or tricyclic antidepressant up to7 days or 5 half-lives (whichever is longer) prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
7. Use of Monoamine oxiadse inhibitors drugs up to 14 days prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
8. History of hepatitis
9. Elevated aspartate aminotransferase/alanine aminotransferase/bilirubin,
10. HIV
11. Excessive use of alcohol/tobacco/caffeine
12. Less than 18 years of age.
13. Has previously received study drug.
14. Has a history of abuse of controlled substances, nasal or otherwise, or has damage to the nasal space, that in the opinion of the investigator might interfere with the ability to absorb RX0041-002.
15. Has severely traumatized mucosa or sepsis in the nasal cavity.
16. Has participated in an investigational study or received an investigational drug within 30 days preceding the randomization.
17. Is a pregnant or nursing mother.
18. Has a positive pregnancy test at Screening or Day -1.
19. Has a history of seizure, with the exception of febrile seizures.
20. Has symptomatic cardiovascular disease, moderate to severe hypertension.
21. Has a known personal or family history of hereditary pseudocholinesterase deficiency. Study participants will be screened by asking about personal or family history of anesthetic reaction, anesthetic death, and previous diagnosis of psuedocholinesterase deficiency in a relative or personally. Subjects identified with pseudocholinesterase deficiency are at risk for delayed recovery with certain anesthetics (e.g. succinylcholine and ester-based anesthetics).
22. Has a known personal or family history of pheochromocytoma. Study participants will be specifically asked if they have been treated for a pheochromocytoma previously or if they have a family member who has been diagnosed with pheochromocytoma (since 10% of these are familial).
23. Has a known personal or family history of adrenal tumor.
24. Clinically significant ECG abnormalities, based upon the impression of the investigator.
25. Has a positive urine test result for drugs of abuse (amphetamines, barbiturates, cocaine metabolites, opiates and oxycodone) or cannabinoids at Screening or on Day 1.
26. Blood chemistry values judged clinically significant by the investigator. aa. Donation of blood (one pint or greater) within four weeks prior to administration of study medication.

bb.Use or intended use of any drug or other product that inhibits or induces cytochrome P450 (CYP) 3A4 within 14 days prior to or during the conduct of the study.

cc.Taking drugs or natural herbal supplements (including St. John'sWort) with known interactions with CYP or with the study drug.

dd.Has consumed or is unwilling to refrain from consumption of foods containing grapefruit, pomelo or Seville oranges from within 7 days prior to Day 1 until end of study.

ee.Not suitable for entry into the study in the opinion of the investigator.

Note: A one-time retest is permitted for any blood test if the original sample was hemolyzed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 32 Hours
Area under the plasma concentration versus time curve (AUC) | 32 Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Clinical Researc, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided